CLINICAL TRIAL: NCT04227223
Title: Oxidative- Antioxidative Balance and Cognitive Functions During Opioid Therapy
Brief Title: Oxidative Balance in Opioid Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R-I-002/307/2019
Record Dates: First submitted 2019-12-29; First posted 2020-01-13 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Pain; Opioids
Keywords: neurological condition; opioids; oxidative balance; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The serum measurements were performed in total group of 50 adult patients: Study Group - 36 patients with chronic Low-Back Pain with opioids pharmacotherapy and Control Group - 14 patients, healthy volunteers. I
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Study Group - 36 patients with chronic Low-Back Pain with opioids pharmacotherapy
  Interventions: Diagnostic Test: biochemical measurements
- Control Group (Active Comparator): Control Group - 14 patients, healthy volunteers.
  Interventions: Diagnostic Test: biochemical measurements

INTERVENTIONS:
Diagnostic Test: biochemical measurements — TOC,TAC, and BDNF measurements are performed using ImAnOx , PerOx and BDNF tests (Immundiagnostik, Germany)

SUMMARY:
The oxidative - antioxidative balance is the crucial mechanism of opioid-induced immunomodulation. Additionally, impairement of cognitive function during opioid therapy is another important side- effect. This phenomenon was clearly described in opioids abuse. This is interesting to evaluate the importance of this subjects in chronic pain patients. The aim of the study was to investigate the oxidative - antioxidative homeostasis and cognitive functions using serum total oxidative capacity (TOC) and total antioxidative capacity (TAC) tests and Brain Derivered Neutrophic Factor (BDNF) in patient with chronic non-cancer pain treated with opioids.

DETAILED DESCRIPTION:
The project was approved in Ethical Committee and supported by Medical University of Bialystok (Poland). The serum TOC and TAC measurements were performed in total group of 50 adult patients: Study Group - 36 patients with chronic Low-Back Pain with opioids pharmacotherapy and Control Group - 14 patients, healthy volunteers. In Study Group anthropometric parameters, duration in opioid therapy, type of opioid, total dose, and form of application were registered.TOC, TAC, and BDNF measurements were performed using ImAnOx, PerOx, BDNF tests (Immundiagnostik, Germany).Data were analyzed using non-parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* minimally, 6 months opioid therapy in chronic Low- Back Pain

Exclusion Criteria:

* depression, steroids- local or systemic administration

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
oxidative balance | 6 months of opioids therapy
  measurements of total oxidative capacity and total antioxidative capacity
cognitive state | 6 months of opioids therapy
  measurements of Brain-derived Neurotrophic Function

CONTACTS AND LOCATIONS:
Overall Officials: Urszula Kosciuczuk, Principal Investigator — Medical University in Bialystok
Locations (1):
- Urszula Kosciuczuk, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: No